CLINICAL TRIAL: NCT05559008
Title: A Umbrella Study in Relapsed/Refractory Peripheral T-cell Lymphoma Guided by Molecular Subtypes
Brief Title: A Umbrella Study in R/R PTCL Guided by Molecular Subtypes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-IIT-umbrella
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Azacitidine; Dasatinib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T1 subtypes based on next generation sequencing results (Experimental): T1 subtypes based on next generation sequencing results
  Interventions: Drug: Azacitidine Injection; Drug: Dasatinib
- T2 subtypes based on next generation sequencing results (Experimental): T2 subtypes based on next generation sequencing results
  Interventions: Drug: Azacitidine Injection; Drug: Linperlisib
- T3.1 subtypes based on next generation sequencing results (Experimental): T3.1 subtypes based on next generation sequencing results
  Interventions: Drug: Tucidinostat; Drug: SHR2554
- T3.2 subtypes based on next generation sequencing results (Experimental): T3.2 subtypes based on next generation sequencing results
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Azacitidine Injection — Azacitidine Injection，SC and Dasatinib PO will be administered in T1 subtypes
  Arms: T1 subtypes based on next generation sequencing results; T2 subtypes based on next generation sequencing results
Drug: Dasatinib — Azacitidine Injection，SC and Dasatinib PO will be administered in T1 subtypes
  Arms: T1 subtypes based on next generation sequencing results
Drug: Linperlisib — Azacitidine Injection，SC and Linperlisib PO will be administered in T2 subtypes
  Arms: T2 subtypes based on next generation sequencing results
Drug: Tucidinostat — Tucidinostat PO and SHR2554 PO will be administered in T3.1 subtypes
  Arms: T3.1 subtypes based on next generation sequencing results
Drug: SHR2554 — Tucidinostat PO and SHR2554 PO will be administered in T3.1 subtypes
  Arms: T3.1 subtypes based on next generation sequencing results
Drug: Camrelizumab — Camrelizumab and Apatinib will be administered in T3.2 subtypes
  Arms: T3.2 subtypes based on next generation sequencing results
Drug: Apatinib — Camrelizumab and Apatinib will be administered in T3.2 subtypes
  Arms: T3.2 subtypes based on next generation sequencing results

SUMMARY:
This is a multicenter, prospective, open-label, interventional umbrella study to evaluate the efficacy and safety of targeted therapies guided by molecular subtypes in patients with relasped or refractory peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed Peripheral T-cell lymphoma (without central nervous system involvement)
2. Relapsed or refractory disease after first line treatment
3. Availability of archival or freshly collected tumor tissue before study enrollment
4. Evaluable lesion by PET-CT or CT scan
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
6. Life expectancy greater than or equal to (>/=) 3 months
7. Informed consent

Exclusion Criteria:

1. Patients with central nervous system (CNS) lymphoma
2. History of malignancies except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
3. Uncontrolled cardio- and cerebro-vascular disease, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
4. Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

   Neutrophils<1.0×10^9/L Platelets<75×10^9/L (Platelets<50×10^9/L in case of bone marrow involvement) ALT or AST is 2.5 times higher than the upper limits of normal (ULN), AKP and bilirubin are 1.5 times higher than the ULN.

   Creatinine is 1.5 times higher than the ULN.
5. HIV-infected patients
6. Active hepatitis infection
7. Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
8. Pregnant or lactation
9. Other medical conditions determined by the researchers that may affect the study For T3.2 should exclude patiens with active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6）(each cycle is 28 days)
  Percentage of participants with complete and partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Complete response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6）(each cycle is 28 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
Duration of response | Baseline up to data cut-off (up to approximately 2 years)
  Duration of response was defined as the time from the date of favorable response until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No